CLINICAL TRIAL: NCT06009705
Title: Efficacy and Safety of Toripalimab Combined With Radiotherapy and S-1 Followed by Adjuvant Toripalimab Maintenance Therapy for Older Patients With Esophageal Cancer
Brief Title: Toripalimab Combined With Radiotherapy and S-1 for Older Patients With Esophageal Cancer
Acronym: Best-EEC
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Best-EEC
Record Dates: First submitted 2023-08-10; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Carcinoma
Keywords: esophageal carcinoma; esophageal cancer; immunotherapy; chemoradiotherapy; toripalimab
MeSH Terms: conditions — Esophageal Neoplasms | interventions — toripalimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: toripalimab — JS001, the active ingredient of toripalimab injection, independently developed by Shanghai Junshi Biomedical Technology Co., Ltd, is an independently developed novel recombinant humanised (degree of 97%) anti-PD-1 monoclonal antibody (Chinese Patent License No. CN104250302B, PCT Patent Publication No. WO2014/206107A1), belonging to the human IgG4/Kappa subtype, and introducing a point mutation at the Serine to Proline (S228P) protein site 228 in the hinge region of the IgG4 heavy chain.

SUMMARY:
This trial aims to assess efficacy and safety of toripalimab combined with radiotherapy and S-1 followed by adjuvant toripalimab maintenance therapy for older patients with stage II-III esophageal cancer.

DETAILED DESCRIPTION:
With the aging of the population, the number of elderly esophageal cancer patients is gradually increasing. For non-metastatic esophageal cancer patients, surgery is the first choice of treatment, but elderly esophageal cancer patients are often unable to tolerate surgical treatment due to more comorbidities and poor physical condition, etc. The results of previous studies have shown that the effect of radiotherapy treatment is also unsatisfactory, and the 5-year survival rate of esophageal cancer patients treated with radiotherapy is only 15-25%, which makes the clinical treatment of elderly patients even more difficult due to their poor physical tolerance. A multicentre randomised phase III clinical trial (NCT02813967) demonstrated that concurrent radiotherapy and S-1 treatment in elderly patients with esophageal cancer was tolerable and provided significant benefit compared with radiotherapy alone. In recent years, tumor immunotherapy has shown some efficacy in the field of cancer treatment by activating the body's own immune system to fight tumors. Therefore, this trial aims to assess efficacy and safety of toripalimab combined with radiotherapy and S-1 followed by adjuvant toripalimab maintenance therapy for older patients with stage II-III esophageal cancer. The primary study endpoints are objective remission rate (ORR), disease control rate (DCR), duration of remission (DOR) and safety. Secondary study endpoints are overall survival (OS) and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written signed informed consent;
* Age ≥65 years old, gender is not limited;
* Histologically or cytologically confirmed esophageal cancer;
* Elderly patients with stage I-III esophageal cancer who are inoperable or refuse to undergo surgery and can tolerate immunotherapy combined with S-1 and radiotherapy;
* Physical status score ECOG 0-2;
* Expected survival ≥ 6 months;
* no serious abnormalities of haematopoietic, cardiac, pulmonary, hepatic and renal functions and immunodeficiency (Haematology: white blood cells ≥3.5×109/L; neutrophils ≥1.5×109/L; haemoglobin ≥90g/L; platelets ≥100×109/L. Liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) ≤2.5 times the upper limit of normal; creatinine ≤1.5 times the upper limit of normal; albumin ≥30 g/L. Coagulation: International Normalised Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, PT or INR is acceptable as long as the PT or INR is within the range of the anticoagulant drug formulation. Echocardiographic assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%). Pulmonary function FEV1 ≥70% of % of predicted value and DLCO ≥60% of % of predicted value).
* Have at least one measurable lesion as judged by RECIST 1.1 criteria.

Exclusion Criteria:

* Distant organ metastases (excluding supraclavicular lymph nodes) as determined by CT evaluation during screening and prior imaging;
* Pre-treatment with oesophageal fistula, perforation, or malignant disease;
* have received prior radiotherapy to the chest;
* having any active autoimmune disease or a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included if hormone replacement therapy is effective), etc.), and a history of immunosuppressive drug use within 28 days, with the exception of the use of hormones for the purpose of dealing with toxicity from radiotherapy;
* Previously received or are receiving other PD-1 antibody therapy or other immunotherapy targeting PD-1/PD-L1, or are currently participating in other interventional clinical studies for treatment;
* Have received other anti-tumour therapy (including herbal therapy with anti-tumour effect) within 4 weeks prior to the first dose of the study; have received long-term systemic immunotherapy or hormone therapy (except physiological replacement therapy, e.g., oral thyroxine for hypothyroidism) within 4 weeks prior to the first dose of the study; and have been treated with other experimental drugs or interventional clinical studies within 4 weeks prior to the first dose of the study;
* Known hypersensitivity to large protein preparations, or to any of the components within toripalimab, S-1 capsules and their preparations;
* Patients with uncontrolled clinical cardiac symptoms or disease such as (1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* with congenital or acquired immune function defects (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥104 copies/ml) or hepatitis C (hepatitis C antibody-positive with HCV-RNA above the lower limit of detection of the analytical method), or active tuberculosis;
* Have an active infection or unexplained fever >38.5°C within 2 weeks prior to screening (at the investigator's discretion, subjects may be enrolled for fever arising from tumours);
* History of malignancy other than oesophageal cancer within the past 5 years, except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix;
* In the judgement of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study in the middle of the study, e.g., suffering from other serious illnesses (including psychiatric illnesses) that require comorbid treatment, family or social factors that may affect the safety of the subject or the collection of trial data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older esophageal cancer patients who receive toripalimab combined with radiotherapy and S-1 followed by adjuvant toripalimab maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of objective remission rate (ORR) in elderly esophageal cancer patients treated with toripalimab in combination with S-1 and radiotherapy. | 2022/10/1-2026/4/30
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Objective remission rate (ORR): defined as the proportion of subjects whose tumor volume shrinks to a pre-specified value and can be maintained for the minimum time frame required, incorporating cases in complete remission (CR) and partial remission (PR).
Assessment of disease control rate (DCR) in elderly esophageal cancer patients treated with toripalimab in combination with S-1 and radiotherapy. | 2022/10/1-2026/4/30
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Disease control rate (DCR): the proportion of patients whose tumors shrank or were stable and remained so for a certain period of time, including complete remission (CR), partial remission (PR) and stable disease (SD).
Assessment of duration of remission (DOR) in elderly esophageal cancer patients treated with toripalimab in combination with S-1 and radiotherapy. | 2022/10/1-2026/4/30
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Duration of remission (DOR): refers to the time between the start of the first assessment of the tumor as complete remission (CR) or partial remission (PR) and the first assessment of PD or death from any cause.
Assessment of the incidence of treatment-related adverse events Incidence of Treatment-Emergent Adverse Events. | 2022/10/1-2026/4/30
  Adverse events are observed during the course of the study and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

SECONDARY OUTCOMES:
Assessment of overall survival (OS) in elderly esophageal cancer patients treated with toripalimab in combination with S-1 and radiotherapy. | 2022/10/1-2026/4/30
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). OS is defined as the time from the start of enrollment to death from any cause.
Assessment of progression-free survival (PFS) in elderly esophageal cancer patients treated with toripalimab in combination with S-1 and radiotherapy. | 2022/10/1-2026/4/30
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). PFS is defined as the time from the start of enrollment until tumor progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Shen, PhD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China